CLINICAL TRIAL: NCT00011791
Title: Catecholamine Reserve and Exercise Tolerance in Subjects With Congenital Adrenal Hyperplasia and Healthy Controls
Brief Title: Catecholamine Reserve and Exercise Tolerance in Healthy Volunteers and Patients With Congenital Adrenal Hyperplasia
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010096; 01-CH-0096
Record Dates: First submitted 2001-02-28; First posted 2001-03-01 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-05-10

CONDITIONS: Congenital Adrenal Hyperplasia; Healthy
Keywords: CAH; Catecholamines; Adrenal Medulla; Endocrine; Congenital Adrenal Hyperplasia; Exercise; Healthy Volunteer
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Motor Activity

SUMMARY:
This study will examine and compare the effects of intense exercise on the release of catecholamines in patients with congenital adrenal hyperplasia (CAH) and in healthy persons. Catecholamines are hormones (adrenaline and noradrenaline) that are produced by the adrenal glands and released into the blood stream during stress, such as trauma, illness, intense exercise, or low blood sugar. The study will also assess exercise tolerance in patients with CAH, compared with healthy persons.

Patients with CAH between the ages of 10 and 40 years who are managing well on standard treatment (glucocorticoids, mineralocorticoids) may be eligible for this study. Healthy volunteers that match the enrolled patients in age, sex, race and body fat will be recruited as control subjects. All candidates will be screened with a medical history, physical examination and electrocardiogram (EKG). Body fat will be measured using an instrument called a Bod Pod. The body fat measurement has two parts: first, the subject sits quietly in a large egg-shaped capsule for about 2 to 3 minutes; then the subject breathes into a plastic tube for one minute, followed by three quick panting breaths. Women will have a urine pregnancy test; pregnant women cannot participate in the study.

Participants will undergo three exercise sessions on separate consecutive mornings after fasting overnight. Before each test, patients (not healthy volunteers) will take either an additional morning dose of hydrocortisone or a placebo (a lookalike pill with no active ingredient). Before each test a thin catheter (plastic tube) will be placed into an arm vein through a needle. A numbing cream can be applied to make the needle stick hurt less. Blood will be drawn through this intravenous (IV) line before, during and after the exercise tests. The first test is a maximal exercise test to determine the individual's maximum exercise fitness capacity. The second two and third tests are a standardized exercise tests. Before the two standardized tests, patients (not healthy volunteers) will take either an additional morning dose of hydrocortisone or a placebo (a lookalike pill with no active ingredient). All tests are done on a stationary bicycle.

Maximal Exercise Test - The subject pedals on a stationary bicycle for about 10 minutes. After a 3-minute warm-up, the workload is increased continuously until either the subject can no longer continue or the physician stops the test for medical reasons. During the exercise, heart rate and heart activity are monitored with an EKG, and the subject wears a nose clip and mouthpiece connected to a breathing tube to measure oxygen use. Blood is drawn before and during the test, totaling no more than 2 tablespoons.

Standardized Exercise Test - The subject pedals on a stationary bicycle for 20 minutes, while wearing the nose clip and mouthpiece to measure oxygen use. For the first 5 minutes, the subject pedals at a speed that elicits 50 percent of maximal effort (determined by the maximal exercise test); the next 10 minutes are at 70 percent of maximal effort; and the last 5 minutes are at 90 percent. Blood samples drawn before, during (at 15 and 20 minutes) and after exercise (at 30, 40 and 60 minutes) total less than 1/2 cup. Heart rate and heart activity are monitored during the test with an EKG, and temperature is measured before and at the end of the test.

DETAILED DESCRIPTION:
Congenital adrenal hyperplasia (CAH) denotes a family of inherited disorders with defects in the cortisol biosynthesis. CAH has been traditionally considered a disease restricted to the adrenal cortex. However, recently observed abnormal adrenomedullary structures in three adrenalectomized patients with classic CAH, as well as low baseline urinary and plasma epinephrine levels in children with CAH suggest that this condition is associated with marked morphological and functional abnormalities of the adrenal medulla.

The adrenal medulla synthesizes and secretes catecholamines, mainly epinephrine. Catecholamines influence virtually all tissues. Yet, the clinical implications of epinephrine deficiency in humans are not clear.

Short-term intense exercise is a natural, quantifiable stimulus of the adrenal cortex and medulla as well as of the sympathetic nervous system. We would like to employ a standard cycle ergometer exercise protocol to study the adrenomedullary and systemic sympathetic function of patients with CAH. This protocol has been run by the Clinical Center Rehabilitation Medicine Department (RMD) for 10 years. No serious adverse effects have been observed or reported in adults and children with a healthy cardiovascular system.

The goal of this protocol is to evaluate adrenomedullary and systemic sympathetic function and exercise tolerance in patients with CAH and in appropriately matched healthy controls using the above standardized cycle ergometer test. Subjects with CAH will exercise with and without doubling their morning dose of hydrocortisone to evaluate whether impairments - if present - can be corrected by a "stress dose" of hydrocortisone. We hypothesize that subjects with CAH have a reduced epinephrine reserve and impaired exercise tolerance, which can at least partially, be corrected by an increase in exogenous hydrocortisone. We will also determine whether the systemic sympathetic nervous system compensates for the adrenomedullary deficiency as observed in states of acquired adrenal insufficiency. The results of this study will increase the understanding of the physiologic interactions between adrenal cortex and adrenal medulla.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age: 9-40 years.

CAH patients on conventional therapy (glucocorticoids, mineralocorticoids) in good clinical management as defined by the following criteria:

1. 17-OH-progesterone level between 100 and 1500 ng/dL;
2. Plasma renin activity normal;
3. Growth rate within 2 SD for age (children);
4. No new signs or symptoms of virilization (clitoral growth, voice deepening) for females.

Healthy volunteers will be matched for age, sex, race and body fat.

EXCLUSION CRITERIA:

Inability to understand or comply with instructions related to the study (as judged by investigator).

Chronic medical conditions other than congenital adrenal hyperplasia except mild conditions (e.g. allergic rhinitis, migraine headaches) will be excluded provided the subjects are not acutely ill and do not require medication for this condition during the study.

Acute medical conditions including intercurrent infection and fever in the preceding 7 days.

Positive pregnancy test.

CAH patients on flutamide.

Tylenol or other acetaminophen-containing medicines (e.g. over-the-counter cold medicines) within 5 days before each test period.

Caffeine, alcohol or strenuous exercise within 24 h before each test period.

Current smokers.

Ages: 9 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2001-02-22; Study Completion 2011-05-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Albert CM, Mittleman MA, Chae CU, Lee IM, Hennekens CH, Manson JE. Triggering of sudden death from cardiac causes by vigorous exertion. N Engl J Med. 2000 Nov 9;343(19):1355-61. doi: 10.1056/NEJM200011093431902. PMID 11070099
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Axelrod J, Reisine TD. Stress hormones: their interaction and regulation. Science. 1984 May 4;224(4648):452-9. doi: 10.1126/science.6143403.